CLINICAL TRIAL: NCT05286697
Title: The Effect of Optic Nerve Diameter on Postoperative Cognitive Function in Patients in Long Trendelenburg Position in Laparoscopic Hysterectomy Surgery
Brief Title: The Effect of Optic Nerve Diameter on Postoperative Cognitive Function in Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09.2021.1035
Record Dates: First submitted 2022-02-22; First posted 2022-03-18 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Intracranial Pressure Increase; Postoperative Cognitive Dysfunction
Keywords: laparoscopic hysterectomy; trendelenburg position; optic nerve sheath diameter (ONSD); Mini Mental State Examination (MMSE); postoperative cognitive dysfunction
MeSH Terms: conditions — Intracranial Hypertension; Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effect of increase intracranial pressure on postoperatve cognitive function (Other): All patient will be given a mini mental test before and after the surgery and the optic nerve diameter will be measured 5 times during the surgery.
  Interventions: Diagnostic Test: measuring optic nerve diameter

INTERVENTIONS:
Diagnostic Test: measuring optic nerve diameter — During the measurement of the optic nerve diameter, a layer of sterile water-soluble gel will be applied on the closed eyelid with a linear 10-5 MHz ultrasound probe.

SUMMARY:
Prospective study, 40 patients ASA 2-3, 30-75 years old who were planned for laparoscopic hysterectomy operation will be included.One day before the operation and postoperative 1.3.7. A mini mental assessment test will be performed on these days.Standard monitoring and Near-Infrared Spectroscopy monitoring to measure cerebral oxygen saturation will be performed on the patients.NIRS sensors will be placed on the right and left sides of the forehead, 2 cm above the eyebrow, before induction of anesthesia. Before the induction of anesthesia, the measurement will begin and the FiO2 (fraction of inspiration oxygen) will be kept at 60%.General anesthesia induction will be made with propofol 2mg/kg, remifentanil 0.5 µg/kg and rocuronium 0.6mg/kg, and maintenance will be provided with 2% sevoflurane.The patient will be intubated and ventilation support will be provided so that the tidal volume is 6-8 ml/kg and the end tidal CO2 is 30-40 mmHg. PEEP (Positive end expiratory pressure) will not be applied to any patient. Intra-abdominal pressure will be maintained at 15 mmHg. All patients will be given 1gr paracetamol and 100mg tramadol for postoperative analgesia.During the measurement of optic nerve diameter, a layer of sterile water-soluble gel will be applied on the closed eyelid with a linear 10-5 MHz ultrasound probe. In our study, ONSDs of all patients will be measured by the same experienced anesthetist. Measurements will be made at 5 different times. 5 minutes after induction of anesthesia in the supine position (T0), 5 minutes after the onset of pneumoperitoneum (T1), 5 minutes after the upright trendelenburg position (T2), at the 2nd hour of the trendelenburg position (T3) and 5 minutes after returning to the supine position at the end of the surgery (T4) .ONSD measurements of the patients measured at 5 different times, peroperative NIRS values, peroperative SpO2, mean blood pressure, peak heart rate, anesthesia time, surgery time, time to stay in the trendelenburg position, partial oxygen saturation (PaO2), PCO2, end-tidal carbon dioxide (ETCO2) and peak airway pressure (pPEAK) will be recorded.

DETAILED DESCRIPTION:
To show whether the relationship between increased intracranial pressure and optic nerve diameter after long (> 2.5 hours) Trendelenburg laparoscopic hysterectomies has an effect on postoperative cognitive functions.

Laparoscopic surgery has been developing rapidly in recent years. The fact that the bleeding risk and hospital stay are less, less pain, faster return to normal work, better cosmetic results and superior patient morbidity have made laparoscopic interventions more preferable (1). CO2 pneumoperitoneum and upright upside-down position (Trendelenburg position) are applied to patients who will undergo laparoscopic surgery for better visualization of the surgical field. However, the combined use of the pneumoperitoneum and trendelenburg position causes an increase in intraabdominal pressure, which triggers many systemic physiological changes, along with a decrease in venous return, and increases cerebral blood flow, intracranial pressure, and intraocular pressure (2,3).

Optic nerve sheath diameter (ONSD), determined by non-invasive ocular sonography, is a simple and reliable method that is an indicator of increased intracranial pressure (ICP) in patients (4). Studies have found 100% sensitivity and specificity in the prediction that if ONSD is >5.5, ICP will be >20 mmHg (5,6).

The effect of ONSD on postoperative delirium or postoperative cognitive dysfunction has not been fully explained in the literature. The aim of our study; To show whether the relationship between increased intracranial pressure and ONSD after long-lasting (>2.5 hours) Trendelenburg laparoscopic hysterectomies has an effect on postoperative cognitive functions.

In this prospective and observational study, 40 patients ASA 2-3, 30-75 years old who were planned for laparoscopic hysterectomy operation will be included. Patients with a previous history of ocular disease, ocular surgery, neurological disease and transient ischemic attack will be excluded from the study. Cases returning to open surgery will be excluded from the study. One day before the operation and postoperative 1.3.7. A mini mental assessment test (MMSE-Mini Mental State Examination) will be performed on these days.

Standard monitoring (electrocardiography-ECG, pulse oximetry, noninvasive arterial blood pressure) and Near-Infrared Spectroscopy (NIRS) monitoring to measure cerebral oxygen saturation will be performed on the patients. NIRS sensors will be placed on the right and left sides of the forehead, 2 cm above the eyebrow, before induction of anesthesia. Before the induction of anesthesia, the measurement will begin and the FiO2 (fraction of inspiration oxygen) will be kept at 60%. If cerebral oxygen decreases by more than 20% or is below 50% absolute, position will be changed or FiO2 will be increased.

General anesthesia induction will be made with propofol 2mg/kg, remifentanil 0.5 µg/kg and rocuronium 0.6mg/kg, and maintenance will be provided with 2% sevoflurane. The patient will be intubated and ventilation support will be provided so that the tidal volume is 6-8 ml/kg and the end tidal CO2 is 30-40 mmHg. PEEP (Positive end expiratory pressure) will not be applied to any patient. Intra-abdominal pressure will be maintained at 15 mmHg. All patients will be given 1gr paracetamol and 100mg tramadol for postoperative analgesia.

During the measurement of optic nerve diameter, a layer of sterile water-soluble gel will be applied on the closed eyelid with a linear 10-5 MHz ultrasound probe. In our study, ONSDs of all patients will be measured by the same experienced anesthetist.

SPSS 21.0 computer program will be used for statistical analysis. Based on our pilot study data, a minimum sample size of 23 patients with 0.05 alpha and 90% power indicated that a sample size would be required.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2-3,
* Patients aged 30-75 years who are scheduled for laparoscopic hysterectomy will be included.

Exclusion Criteria:

* Patients with a previous history of ocular disease,
* undergoing ocular surgery,
* patients with neurological disease and transient ischemic attack,
* Cases who converted to open surgery will be excluded from the study.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Optic nerve diameter measurement | Intraoperative
  all patients' Optic nerve diameter will be measured by the same experienced anesthetist and recorded

SECONDARY OUTCOMES:
mini mental test | Baseline (before surgery) and immediately after surgery.
  mini mental assessment test will be done and recorded for the patients.

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No